CLINICAL TRIAL: NCT06778265
Title: An Exploratory Clinical Study to Evaluate UX-DA001 Injection (Human Midbrain Dopaminergic Progenitor Cells Injection) in Subjects With Idiopathic Parkinson's Disease
Brief Title: An Exploratory Clinical Study of UX-DA001 in Subjects With Idiopathic Parkinson's Disease
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai UniXell Biotechnology Co., Ltd (Industry)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX-DA001-101
Record Dates: First submitted 2024-12-30; First posted 2025-01-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: Idiopathic Parkinson´s Disease; autologous iPSC derived mDAPs; Midbrain Dopaminergic Progenitors; Induced pluripotent stem cells; mDAPs; stem cells; iPSC derived product
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: open-label, multi-center, dose-escalation and dose-expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UX-DA001 (Experimental)
  Interventions: Biological: UX-DA001

INTERVENTIONS:
Biological: UX-DA001 — UX-DA001 (Human Midbrain Dopaminergic Progenitor Cells) is used for treating patients with iPD via implanting into bilateral putamina under stereotactic neurosurgery.
  Two dose levels will be planned. Each patient only receives one corresponding dose of UX-DA001.

SUMMARY:
This clinical study is designed to explore the safety and tolerability of UX-DA001. It will also explore if UX-DA001 works to improve motor function in subjects with Parkinson's disease. UX-DA001 manufactured from participant's own cells will differentiate into mature dopaminergic neurons after being transplanted into the brain of the participant.

DETAILED DESCRIPTION:
This study is an open-label, multi-center, dose-escalation and dose-expansion exploratory clinical study to evaluate the safety, tolerability, and potential efficacy of UX-DA001 Injection at different dose levels implanted in subjects with idiopathic PD.

Each subject receives only one dose of UX-DA001 for implantation into the putamen bilaterally using stereotactic neurosurgery under general anesthesia. Safety and tolerability of UX-DA001 and its effect on Parkinson's disease symptoms are assessed for 2 years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects or their legally acceptable representative understand and comply with the study procedures, agree to participate in the clinical trial, and sign the ICF;
2. Aged between 50-75 years old, male or female;
3. Subjects diagnosed with idiopathic PD, with a medical history of 5-20 years;
4. Having received standard anti-PD treatment and been given optimal anti-PD treatment under the guidance of the investigator, but the efficacy has significantly declined;
5. Good response to levodopa medications; the LCT shows that the maximum improvement rate of the UPDRS part III score exceeds 30%;
6. The modified H&Y scale of clinical "OFF" period is ≥ Stage 3 and ≤ Stage 4;
7. Taking a stable dosage of anti-PD medications for at least 4 weeks;
8. Good physical condition or stable concomitant diseases;
9. With reliable caregivers who can cooperate to complete the assessment items;
10. Subjects with good compliance.

Exclusion Criteria:

1. PD Subjects in whom previous genetic testing has found a GBA gene mutation or PD Subjects whom the investigator considers unsuitable for participation in this clinical study due to other gene mutations;
2. Subjects with the atypical Parkinson's syndrome or secondary Parkinson's syndrome;
3. Subjects with HIV, HBV, HCV, treponema pallidum (TP) infection, or other active infections;
4. Subjects infected with HTLV, EBV or CMV whose infection renders their blood cells unsuitable for cell product preparation;
5. Subjects with a known hereditary disorder;
6. Subjects with any history of malignancy;
7. Subjects with other serious systemic diseases or functional disorders;
8. Accompanied by other serious central nervous system diseases or serious cognitive and mental disorders;
9. Subjects who are currently receiving or have previously received cell therapy or other medicine effecting safety and efficacy assessement;
10. Subjects whose prior head CT/MRI examinations indicate brain injury, or Subjects with imaging abnormalities in the striatum and other brain regions leading to a significant increase in surgical risk, or Subjects who have previously undergone brain surgery;
11. Subjects with clinically significant abnormal results in coagulation function, or Subjects who have been using anticoagulants for a long time and cannot discontinue use;
12. Subjects with a history of severe allergy or hypersensitivity reactions, or a known history of hypersensitivity, or a history of intolerance to the investigational cellular drug or its excipients;
13. Subjects who have undergone other surgeries within the past six months that the investigator deems may affect this trial, or Subjects who cannot tolerate general anesthesia or stereotactic surgery;
14. Subjects with contraindications to MRI and PET scans;
15. Subjects with a history of alcoholism or drug abuse;
16. Women during pregnancy or lactation;
17. Subjects who have participated in other interventional clinical trials or similar clinical trials within the past 3 months;
18. Subjects with other conditions that are not suitable for participation in the clinical study as judged by the investigator.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and and severity of adverse events (AEs) associated with surgery and/or investigational product | within 4 weeks post surgery
  The incidence and and severity of adverse events (AEs) associated with surgery and/or investigational product during the surgical treatment period and the 4-week postoperative observation period.
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
The incidence and severity of AEs/serious adverse events (SAEs) | From baseline to 2 years post surgery
  The incidence and severity of AEs/serious adverse events (SAEs) during the study, including AEs and SAEs during the surgery treatment period, postoperative observation period, and follow-up period. Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
18F-FP-CIT uptake using positron emission tomography (PET) | From baseline to 2 years post surgery
  Changes in 18F-FP-CIT uptake using positron emission tomography (PET) from baseline.
The situation of implantation and overgrowth of transplanted cells using cranial MRI | From baseline to 2 years post surgery
  Volume changes of transplanted cells using cranial magnetic resonance imaging (MRI)
Changes in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) score, part III, from baseline. | From baseline to 2 years post surgery
  Minimum score: 0; Maximum score: 132; Higher scores mean a worse outcome.
Changes in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) score, part II, from baseline. | From baseline to 2 years post surgery
  Minimum score: 0; Maximum score: 52; Higher scores mean a worse outcome.
Changes in modified modified Hoehn-Yahr (H&Y) scale from baseline | From baseline to 2 years post surgery
  Grade 0~Grade 5, lower grade means a better outcome
Changes in daily levodopa equivalent dose (LED) from baseline. | From baseline to 2 years post surgery
Changes in the scores of non-motor symptom scales (NMSS) from baseline. | From baseline to 2 years post surgery
  Minimum score: 0; Maximum score: 960; Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, MD, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No